CLINICAL TRIAL: NCT02978144
Title: In Vivo Imaging of Destructive Processes in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Lung Imaging of Apoptosis in Chronic Obstructive Pulmonary Disease (COPD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty finding Annexin study drug supplier
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAR0417; 1R01HL131960-01 (NIH)
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Phase 2
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: All study participants will receive study drug Annexin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): All study participants will be administered Annexin (study drug also known as 99mTc-Annexin V-128 (AxV-128/Tc)) intravenously (IV) followed by SPECT-CT imaging scan.
  Interventions: Drug: AxV-128/Tc

INTERVENTIONS:
Drug: AxV-128/Tc — Study drug 99mTc-Annexin V-128 (AxV-128/Tc) is administered intravenously prior to SPECT/CT imaging.

SUMMARY:
This is a prospective interventional study examining the use of Annexin - a radioactive tracer, in assessing lung damage in healthy volunteers, healthy volunteers actively smoking, and patients with moderate and severe chronic obstructive pulmonary disease (COPD). All study participants will undergo a CT scan, pulmonary testing, and blood test. The study procedures are done in one day. The aim of this study is to determine if Annexin can be used as a marker to detect lung injury early on and aid in the future diagnosis of COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the third leading cause of death and is characterized by clinical symptoms and spirometry. Additional measures for diagnosis can be taken using imaging modalities such as CT. However, the evaluation of lung destruction in COPD is limited by the inability to visualize the activation of pathological processes since imaging modalities are only able to evaluate end-organ damage.

In the current study, the investigators aim to assess a molecular imaging probe targeting apoptosis, a cellular process known to be pathogenic in COPD. Apoptosis, a process of programmed cellular death, correlates with COPD severity and is not seen in the normal adult lung. In the past several years the investigators have demonstrated the successful ability of AxV-128/Tc to detect apoptosis in vivo in a preclinical animal model of smoke exposure emphysema model. Additionally, Phase 1 studies have demonstrated safety of this agent in healthy patients. Therefore, the investigators will bring 99mTc-Annexin V-128 (AxV-128/Tc) forward as a probe to image the apoptotic disease process of the lung in patients with COPD. The investigators will determine if the imaging signal correlates with serum biomarkers of apoptosis and inflammation. It is the investigators' hypothesis that AxV-128/99mTc imaging will show increased uptake in the lungs of patients with COPD, and that this signal intensity will correlate with accepted markers of apoptosis and inflammation. If successful, such an approach will be a powerful tool to potentially predict disease progression after diagnosis, identify patients at risk for disease exacerbation related lung function decline, and monitor response to disease targeted therapy.

The total effective dose from the combined single-photon emission computed tomography (SPECT) and computerized tomography (CT) scans is 6.2 millisievert (mSv). This effective dose is below what a patient receives during a standard 2 dose rest and stress cardiac nuclear imaging study and well within the range of current clinical nuclear imaging tests. The exact long term risk for development of cancer from diagnostic radiological procedures is currently under debate but all imaging procedures in this study are aimed to keep total radiation burden As Low As Reasonably Achievable (ALARA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate COPD: Global Initiative for Chronic Obstructive Lung Disease (GOLD) Stage II, forced expiratory volume 1 (FEV1)/forced vital capacity (FVC) < 0.7 and FEV1 50-79% predicted
* Patients with severe COPD: GOLD Stage III-IV, FEV1/FVC < 0.7 and FEV1 < 50% predicted
* Healthy controls who are currently smoking (> 10 pack years) with normal spirometry (FEV1 > 80% and FEV1/FVC > 70%)
* Healthy controls who never smoked (less than 100 lifetime cigarettes) with normal spirometry (FEV1 > 80% and FEV1/FVC > 70%)

Exclusion Criteria:

* Age < 18 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gebhard Wagener, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 34
Completed | 0
Not Completed | 34

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 34
Age, Customized [Count of Participants; unit: Participants]
  18 - 39 years | 0
  40 - 59 years | 14
  60 - 79 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 24
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean AxV-128/Tc Uptake
Description: Mean ± standard deviation (SD) for values for uptake of AxV-128/Tc for individual lobes and for lungs will be determined for each COPD group and compared using unpaired t-test for values with Gaussian distribution and Mann Whitney (Wilcoxon rank) test for continuous variables without normal distribution.
Time Frame: At first visit (Day 1) and if available, at up to 18 months from the initial scan
Population: Data was not collected. Participants were enrolled prior to the study termination but were not administered the study intervention due to inability to obtain a drug supplier.
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 18 months from the initial scan
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT02978144/Prot_SAP_000.pdf